CLINICAL TRIAL: NCT02517476
Title: Effect of Early Nutritional Therapy on Frailty, Functional Outcomes and Recovery of Undernourished Medical Inpatients Trial: The EFFORT Trial
Brief Title: Effect of Early Nutritional Therapy on Frailty, Functional Outcomes and Recovery of Undernourished Medical Inpatients Trial
Acronym: EFFORT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other); Insel Gruppe AG, University Hospital Bern (Other); Luzerner Kantonsspital (Other); Kantonsspital Münsterlingen (Other); Clinical Trial Unit, University Hospital Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Philipp Schuetz, Prof. Dr. med., University Hospital, Basel, Switzerland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EKNZ 2014-001
Record Dates: First submitted 2015-07-30; First posted 2015-08-07 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional support (Experimental): For the purpose of this study, we have developed nutritional guidelines by consensus and adapted to current guidelines (e.g., ESPEN, ASPEN). These guidelines specify a reinforced nutritional therapy strategy to cover nutritional requirements, focusing on nutritional targets based on the specific nutritional diagnoses defined by the IDNT. The nutritional guidelines may vary according to important medical diagnoses (i.e. renal failure). They specify not only nutritional targets, but also escalation of the route (i.e. food fortification, oral, enteral, parenteral) if targets cannot be achieved (≤75%) every 5 hours. Nutritional goals are being assessed daily in patients in the intervention group.
  Interventions: Dietary Supplement: Nutritional therapy
- Usual care ("appetite-guided") controls (No Intervention): In control patients, we will use conventional nutrition according to the ability and desire of the patient to eat, using standard care food provided by the hospital kitchen ("appetite-guided").

INTERVENTIONS:
Dietary Supplement: Nutritional therapy — Any nutritional product and route (i.e. food fortification, oral, enteral, parenteral) is possible to reach goals
  Arms: Nutritional support

SUMMARY:
The aims of the randomized-controlled, multicenter EFFORT trial are to assess the effects of early nutritional therapy in regard to effectiveness, safety and costs when applied to the heterogenous, polymorbid medical inpatient population. EFFORT will not only answer the question about overall benefit or harm, but using a physio-pathological mechanistic approach, it also will explore and provide conclusive answers about whether, why, how, and in which patient populations nutritional therapy does and does not works.

DETAILED DESCRIPTION:
The aims of the randomized-controlled, multicenter EFFORT trial are to test the hypothesis that in medical inpatients at risk for undernutrition defined by the nutritional risk score (NRS 2002), early tailored nutritional therapy to reach nutritional targets based on individualized nutritional counseling is a cost-effective strategy to prevent mortality, morbidity and functional decline.

The primary composite endpoint is combined adverse outcome within 30 days defined as (a) all-cause mortality, (b) admission to the intensive care unit from the medical ward, (c) major complications, (d) unplanned hospital readmissions and (d) decline in functional outcome from admission to day 30 assessed by Barthel's index (-10%). Secondary endpoints include (a) each single component of the primary endpoint (b) short-term nutritional and functional outcomes from inclusion to day 10 or hospital discharge; (c) hospital outcomes; (d) 30-day and 180-day outcomes (e) Other safety endpoints including adverse gastrointestinal effects associated with nutritional therapy assessed daily until hospital discharge.

The investigators will include unselected adult medical inpatients at risk of undernutrition [NRS≥3 points] and an expected hospital stay of ≥5 days who are willing to provide informed consent. The investigators will exclude patients in critical care or post-operative state, unable to swallow, at long-term need for parenteral/enteral nutrition, in terminal condition, pregnant, with acute pancreatitis or acute liver failure, with anorexia nervosa, that were earlier included into the trial Patients in the intervention group will receive individualized nutritional therapy to reach nutritional targets (caloric, protein, micronutrients, other) based on a predefined nutritional strategy. In control patients, according to patients' appetite, standard hospital nutrition will be served. Nutritional therapy may be started in control patients, if any sort of swallowing disorders develops or if patients need to be prepared for operation. All patients will be re-assessed daily during the hospital stay for nutritional intake and nutritional therapy may be escalated every 24-48 hours (food fortification, oral supplements, enteral, parenteral nutrition) if targets are not met (at least 75% of targets).

The targeted sample size is 2000 - 3000 patients. The inclusion of 2000 - 3000 patients will provide between 76% and 91% power to detect a reduction in the primary endpoint of 15% (from 40% to 34%) assuming a lost to follow up rate of 10%.

ELIGIBILITY:
Inclusion criteria:

* NRS ≥3 points
* expected hospital LOS ≥5 days (as estimated by the treating physician team)
* willingness to provide informed consent (see informed consent statement)

Exclusion criteria

* initially admitted to critical care units (except intermediate care)
* scheduled for surgery or in an immediate post-operative state
* unable to ingest oral nutrition and thus need for enteral or parenteral nutrition
* admitted with, or scheduled for, total parenteral nutrition or tube feeding
* currently under nutritional therapy (defined by at least one visit with a dietician in the last month)
* who are hospitalized because of anorexia nervosa
* in terminal condition (end of life situation)
* hospitalized due to acute pancreatitis
* hospitalized due to acute liver failure
* earlier inclusion into this trial
* cystic fibrosis
* patients after gastric bypass operations
* stem cell transplantation
* any contraindication against nutritional therapy (i.e., enteral and/or parenteral)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2088 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
primary composite endpoint | measured at day 30 by telephone interview
  Number of participants with adverse events including
  1. All-cause mortality
  2. Admission to the intensive care unit
  3. Unplanned hospital readmission after hospital discharge
  4. Major complications including nosocomial infection or abscess requiring antibiotic treatment, respiratory failure with need for invasive or non-invasive ventilation, major cardiovascular event or pulmonary embolism, acute renal failure (defined by 2x increase of baseline creatinine or new requirement of dialysis), gastro-intestinal hemorrhage or intestinal perforation assessed by medical chart review and telephone interview
  5. decline in functional status of 10% or more from admission to day 30 measured by the Barthel's index assessed by patient interview on admission and after 30 days

SECONDARY OUTCOMES:
Weight change | measured at day 30 by telephone interview
  change in weight and BMI from inclusion to day 30 by patient interview and medical chart review
lenght of hospital stay | participants will be followed for the duration of hospital stay with an expected average of 10 days
  days in the hospital within index hospitalisation and within the 30 days of follow up measured by patient interview and medical chart review
Improvement in quality of life | measured at days 30 and 180 by telephone interview
  Improvement in quality of life measured with the EuroQol Group 5-Dimension Self-Report Questionnaire on admission and during follow up measured by patient interview
Combined safety endpoints in regard to side effects from nutritional therapy | measured at day 30
  Number of participants with side effects from nutritional therapy including
  (a) adverse gastrointestinal effects (diarrhea, nausea, vomiting, abdominal pain) assessed by patient interview (yes/no) b) Complications due to tube feeding or center catheter for parenteral nutrition assessed by medical chart review (c) Refeeding syndrome assessed by chart review (d) Acute pancreatitis defined as 2 out of 3 criteria: abdominal pain, 3-fold increase in lipase or amylase, characteristic imaging findings assessed by chart review (e) Liver or gall bladder dysfunction assessed by chart review (f) Hyperglycemia (defined as glucose levels >12mmol/l or persistent levels >10mmol/l in patients without diabetes or well controlled diabetes) assessed by medical chart review
new decubital ulcer | assessed on the day of hospital discharge after an expected average of 10 days
  Clinical diagnosis of decubital ulcer with onset after study inclusion measured by patient interview and medical chart review
Discharge location | assessed on the day of hospital discharge after an expected average of 10 days
  proportion discharge home or to a rehab facility measured by patient interview and medical chart review

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Schuetz, Prof. Dr., Principal Investigator — University Clinic, Kantonsspital Aarau
Locations (1):
- University Clinic, Kantonsspital Aarau, Aarau, Canton of Aargau, Switzerland

REFERENCES:
- [Background] Schuetz P. "Eat your lunch!" - controversies in the nutrition of the acutely, non-critically ill medical inpatient. Swiss Med Wkly. 2015 Apr 23;145:w14132. doi: 10.4414/smw.2015.14132. eCollection 2015. PMID 25906253
- [Background] Schutz P, Bally M, Stanga Z, Keller U. Loss of appetite in acutely ill medical inpatients: physiological response or therapeutic target? Swiss Med Wkly. 2014 Apr 29;144:w13957. doi: 10.4414/smw.2014.13957. eCollection 2014. PMID 24782139
- [Derived] Wunderle C, Martin E, Wittig A, Tribolet P, Lutz TA, Koster-Hegmann C, Stanga Z, Mueller B, Schuetz P. Comparison of the inflammatory biomarkers IL- 6, TNF-alpha, and CRP to predict the effect of nutritional therapy on mortality in medical patients at risk of malnutrition : A secondary analysis of the randomized clinical trial EFFORT. J Inflamm (Lond). 2025 Apr 24;22(1):16. doi: 10.1186/s12950-025-00442-0. PMID 40275239
- [Derived] Tribolet P, Wunderle C, Kaegi-Braun N, Buchmueller L, Laager R, Stanga Z, Mueller B, Wagner KH, Schuetz P. Evaluating repeated handgrip strength measurements as predictors of mortality in malnourished hospitalized patients. Secondary analysis of a randomized controlled trial. Eur J Clin Nutr. 2025 Sep;79(9):897-903. doi: 10.1038/s41430-025-01618-w. Epub 2025 Apr 16. PMID 40240521
- [Derived] Diethelm J, Wunderle C, van Zanten ARH, Tribolet P, Stanga Z, Mueller B, Schuetz P. Urea-to-creatinine ratio as a biomarker for clinical outcome and response to nutritional support in non-critically ill patients: A secondary analysis of a randomized controlled trial. Clin Nutr ESPEN. 2025 Jun;67:242-249. doi: 10.1016/j.clnesp.2025.03.042. Epub 2025 Mar 21. PMID 40122337
- [Derived] Randegger S, Wunderle C, Johansen OE, Tribolet P, Pavlicek V, Braendle M, Henzen C, Thomann R, Neyer P, Stanga Z, Mueller B, Schuetz P. Low plasma pancreatic lipase as a novel predictor of nutritional target achievement and response to nutritional interventions in malnourished inpatients: Secondary analysis of a randomized clinical trial. Clin Nutr. 2025 Apr;47:196-203. doi: 10.1016/j.clnu.2025.02.029. Epub 2025 Feb 25. PMID 40037114
- [Derived] Buchmueller LC, Wunderle C, Laager R, Bernasconi L, Neyer PJ, Tribolet P, Stanga Z, Mueller B, Schuetz P. Association of phenylalanine and tyrosine metabolism with mortality and response to nutritional support among patients at nutritional risk: a secondary analysis of the randomized clinical trial EFFORT. Front Nutr. 2024 Nov 12;11:1451081. doi: 10.3389/fnut.2024.1451081. eCollection 2024. PMID 39600719
- [Derived] Wunderle C, Suter SS, Endner N, Haenggi E, Kaegi-Braun N, Tribolet P, Stanga Z, Mueller B, Schuetz P. Sex differences in clinical presentation, treatment response, and side effects of nutritional therapy among patients at nutritional risk: a secondary analysis of the randomized clinical trial EFFORT. Am J Clin Nutr. 2024 Nov;120(5):1225-1232. doi: 10.1016/j.ajcnut.2024.09.020. Epub 2024 Sep 21. PMID 39307186
- [Derived] Wunderle C, Ciobanu C, Ritz J, Tribolet P, Neyer P, Bernasconi L, Stanga Z, Mueller B, Schuetz P. Association of leucine and other branched chain amino acids with clinical outcomes in malnourished inpatients: a secondary analysis of the randomized clinical trial EFFORT. Eur J Clin Nutr. 2025 Jan;79(1):42-49. doi: 10.1038/s41430-024-01507-8. Epub 2024 Sep 8. PMID 39245679
- [Derived] Olpe T, Wunderle C, Bargetzi L, Tribolet P, Laviano A, Stanga Z, Prado CM, Mueller B, Schuetz P. Muscle matters: Prognostic implications of malnutrition and muscle health parameters in patients with cancer. A secondary analysis of a randomised trial. Clin Nutr. 2024 Sep;43(9):2255-2262. doi: 10.1016/j.clnu.2024.07.020. Epub 2024 Aug 2. PMID 39181036
- [Derived] Keller B, Wunderle C, Tribolet P, Stanga Z, Kaegi-Braun N, Mueller B, Schuetz P. Nutritional support in hospitalised patients with diabetes and risk for malnutrition: a secondary analysis of an investigator-initiated, Swiss, randomised controlled multicentre trial. BMJ Open. 2024 Aug 17;14(8):e084754. doi: 10.1136/bmjopen-2024-084754. PMID 39153787
- [Derived] Stumpf F, Wunderle C, Ritz J, Bernasconi L, Neyer P, Tribolet P, Stanga Z, Mueller B, Bischoff SC, Schuetz P. Prognostic implications of the arginine metabolism in patients at nutritional risk: A secondary analysis of the randomized EFFORT trial. Clin Nutr. 2024 Mar;43(3):660-673. doi: 10.1016/j.clnu.2024.01.012. Epub 2024 Jan 22. PMID 38309228
- [Derived] Wunderle C, Siegenthaler J, Seres D, Owen-Michaane M, Tribolet P, Stanga Z, Mueller B, Schuetz P. Adaptation of nutritional risk screening tools may better predict response to nutritional treatment: a secondary analysis of the randomized controlled trial Effect of early nutritional therapy on Frailty, Functional Outcomes, and Recovery of malnourished medical inpatients Trial (EFFORT). Am J Clin Nutr. 2024 Mar;119(3):800-808. doi: 10.1016/j.ajcnut.2024.01.013. Epub 2024 Jan 28. PMID 38290574
- [Derived] Haenggi E, Kaegi-Braun N, Wunderle C, Tribolet P, Mueller B, Stanga Z, Schuetz P. Red blood cell distribution width (RDW) - A new nutritional biomarker to assess nutritional risk and response to nutritional therapy? Clin Nutr. 2024 Feb;43(2):575-585. doi: 10.1016/j.clnu.2024.01.001. Epub 2024 Jan 5. PMID 38242035
- [Derived] Durmisi M, Kaegi-Braun N, Muller NA, Wunderle C, Tribolet P, Stanga Z, Mueller B, Schuetz P. Association of admission cortisol levels with outcomes and treatment response in patients at nutritional risk : A secondary analysis of a randomized clinical trial. Nutr J. 2023 Nov 15;22(1):59. doi: 10.1186/s12937-023-00881-6. PMID 37968689
- [Derived] Boesiger F, Poggioli A, Netzhammer C, Bretscher C, Kaegi-Braun N, Tribolet P, Wunderle C, Kutz A, Lobo DN, Stanga Z, Mueller B, Schuetz P. Changes in serum albumin concentrations over 7 days in medical inpatients with and without nutritional support. A secondary post-hoc analysis of a randomized clinical trial. Eur J Clin Nutr. 2023 Oct;77(10):989-997. doi: 10.1038/s41430-023-01303-w. Epub 2023 Jul 7. PMID 37419969
- [Derived] Baumgartner A, Olpe T, Griot S, Mentil N, Staub N, Burn F, Schindera S, Kaegi-Braun N, Tribolet P, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Association of CT-based diagnosis of sarcopenia with prognosis and treatment response in patients at risk of malnutrition - A secondary analysis of the Effect of early nutritional support on Frailty, Functional Outcomes, and Recovery of malnourished medical inpatients Trial (EFFORT) trial. Clin Nutr. 2023 Feb;42(2):199-207. doi: 10.1016/j.clnu.2022.12.006. Epub 2022 Dec 22. PMID 36603460
- [Derived] Bretscher C, Buergin M, Gurzeler G, Kagi-Braun N, Gressies C, Tribolet P, Lobo DN, Evans DC, Stanga Z, Mueller B, Schuetz P; EFFORT study team. Association between prealbumin, all-cause mortality, and response to nutrition treatment in patients at nutrition risk: Secondary analysis of a randomized controlled trial. JPEN J Parenter Enteral Nutr. 2023 Mar;47(3):408-419. doi: 10.1002/jpen.2470. Epub 2023 Jan 27. PMID 36587281
- [Derived] Stalder L, Kaegi-Braun N, Gressies C, Gregoriano C, Tribolet P, Lobo DN, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Prospective validation of five malnutrition screening and assessment instruments among medical inpatients: Secondary analysis of a randomized clinical trial. Clin Nutr. 2022 Jun;41(6):1307-1315. doi: 10.1016/j.clnu.2022.04.025. Epub 2022 Apr 26. PMID 35552050
- [Derived] Struja T, Laczko E, Wolski W, Schlapbach R, Mueller B, Roschitzki B, Schuetz P. Association of proteomic markers with nutritional risk and response to nutritional support: A secondary pilot study of the EFFORT trial using an untargeted proteomics approach. Clin Nutr ESPEN. 2022 Apr;48:282-290. doi: 10.1016/j.clnesp.2022.01.035. Epub 2022 Feb 2. PMID 35331503
- [Derived] Kaegi-Braun N, Boesiger F, Tribolet P, Gomes F, Kutz A, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Lobo DN, Cederholm T, Mueller B, Schuetz P. Validation of modified GLIM criteria to predict adverse clinical outcome and response to nutritional treatment: A secondary analysis of a randomized clinical trial. Clin Nutr. 2022 Apr;41(4):795-804. doi: 10.1016/j.clnu.2022.02.009. Epub 2022 Feb 17. PMID 35263688
- [Derived] Bretschera C, Boesiger F, Kaegi-Braun N, Hersberger L, Lobo DN, Evans DC, Tribolet P, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Admission serum albumin concentrations and response to nutritional therapy in hospitalised patients at malnutrition risk: Secondary analysis of a randomised clinical trial. EClinicalMedicine. 2022 Feb 11;45:101301. doi: 10.1016/j.eclinm.2022.101301. eCollection 2022 Mar. PMID 35198927
- [Derived] Hersberger L, Dietz A, Burgler H, Bargetzi A, Bargetzi L, Kagi-Braun N, Tribolet P, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Individualized Nutritional Support for Hospitalized Patients With Chronic Heart Failure. J Am Coll Cardiol. 2021 May 11;77(18):2307-2319. doi: 10.1016/j.jacc.2021.03.232. PMID 33958128
- [Derived] Bargetzi A, Emmenegger N, Wildisen S, Nickler M, Bargetzi L, Hersberger L, Segerer S, Kaegi-Braun N, Tribolet P, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Admission kidney function is a strong predictor for the response to nutritional support in patients at nutritional risk. Clin Nutr. 2021 May;40(5):2762-2771. doi: 10.1016/j.clnu.2021.03.013. Epub 2021 Mar 15. PMID 33933742
- [Derived] Kaegi-Braun N, Tribolet P, Baumgartner A, Fehr R, Baechli V, Geiser M, Deiss M, Gomes F, Kutz A, Hoess C, Pavlicek V, Schmid S, Bilz S, Sigrist S, Brandle M, Benz C, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Value of handgrip strength to predict clinical outcomes and therapeutic response in malnourished medical inpatients: Secondary analysis of a randomized controlled trial. Am J Clin Nutr. 2021 Aug 2;114(2):731-740. doi: 10.1093/ajcn/nqab042. PMID 33829236
- [Derived] Baumgartner A, Hasenboehler F, Cantone J, Hersberger L, Bargetzi A, Bargetzi L, Kaegi-Braun N, Tribolet P, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Effect of nutritional support in patients with lower respiratory tract infection: Secondary analysis of a randomized clinical trial. Clin Nutr. 2021 Apr;40(4):1843-1850. doi: 10.1016/j.clnu.2020.10.009. Epub 2020 Oct 10. PMID 33081983
- [Derived] Kaegi-Braun N, Tribolet P, Gomes F, Fehr R, Baechli V, Geiser M, Deiss M, Kutz A, Bregenzer T, Hoess C, Pavlicek V, Schmid S, Bilz S, Sigrist S, Brandle M, Benz C, Henzen C, Mattmann S, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Six-month outcomes after individualized nutritional support during the hospital stay in medical patients at nutritional risk: Secondary analysis of a prospective randomized trial. Clin Nutr. 2021 Mar;40(3):812-819. doi: 10.1016/j.clnu.2020.08.019. Epub 2020 Sep 5. PMID 32919819
- [Derived] Merker M, Felder M, Gueissaz L, Bolliger R, Tribolet P, Kagi-Braun N, Gomes F, Hoess C, Pavlicek V, Bilz S, Sigrist S, Brandle M, Henzen C, Thomann R, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B, Schuetz P. Association of Baseline Inflammation With Effectiveness of Nutritional Support Among Patients With Disease-Related Malnutrition: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2020 Mar 2;3(3):e200663. doi: 10.1001/jamanetworkopen.2020.0663. PMID 32154887
- [Derived] Schuetz P, Sulo S, Walzer S, Vollmer L, Stanga Z, Gomes F, Rueda R, Mueller B, Partridge J; EFFORT trial collaborators. Economic evaluation of individualized nutritional support in medical inpatients: Secondary analysis of the EFFORT trial. Clin Nutr. 2020 Nov;39(11):3361-3368. doi: 10.1016/j.clnu.2020.02.023. Epub 2020 Feb 25. PMID 32147200
- [Derived] Schuetz P, Fehr R, Baechli V, Geiser M, Deiss M, Gomes F, Kutz A, Tribolet P, Bregenzer T, Braun N, Hoess C, Pavlicek V, Schmid S, Bilz S, Sigrist S, Brandle M, Benz C, Henzen C, Mattmann S, Thomann R, Brand C, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B. Individualised nutritional support in medical inpatients at nutritional risk: a randomised clinical trial. Lancet. 2019 Jun 8;393(10188):2312-2321. doi: 10.1016/S0140-6736(18)32776-4. Epub 2019 Apr 25. PMID 31030981